CLINICAL TRIAL: NCT04783571
Title: Effects of Auditory Stimulation on Sleep and Memory in Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dara S. Manoach, PhD, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2018P002573
Record Dates: First submitted 2021-02-19; First posted 2021-03-05 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia
Keywords: sleep; memory; schizophrenia; auditory stimulation
MeSH Terms: conditions — Schizophrenia | interventions — Acoustic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizophrenia (Experimental): Adult outpatients with a diagnosis of schizophrenia.
  Interventions: Other: Placebo; Other: Auditory Stimulation
- Healthy Controls (Experimental): Adult participants screened to exclude a personal history of mental illness, family history of schizophrenia spectrum disorder, and psychoactive medication use.
  Interventions: Other: Placebo; Other: Auditory Stimulation

INTERVENTIONS:
Other: Placebo — Auditory stimulation will not be delivered during the nap
Other: Auditory Stimulation — Auditory stimulation will be delivered during the nap

SUMMARY:
The investigators will test the hypothesis that auditory stimulation (playing quiet sounds during sleep) can normalize brain activity during sleep and improve memory in patients with schizophrenia. The investigators will do this by measuring sleep and memory performance under two conditions separated by one week: receiving auditory stimulation during sleep and not receiving auditory stimulation during sleep. The investigators will study healthy subjects and outpatients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

For healthy controls:

* Male and female subjects
* 18-50 years of age
* Proficient in English

For schizophrenia patients:

* Male and female schizophrenia outpatients
* 18-50 years of age
* Proficient in English
* Able to give informed consent

Exclusion Criteria:

* Pregnant females
* Current use of psychotropic medications (healthy controls only)
* A history of head injury resulting in prolonged loss of consciousness or other neurological sequelae
* IQ <85
* Neurological disorder (including seizure disorder)
* Significant hearing or vision loss
* Current substance abuse or dependence (nicotine abuse or dependence is not exclusionary)
* Any unstable chronic medical condition that affects sleep
* Diagnosed sleep disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in slow-oscillation spindle coupling | Placebo and auditory stimulation naps will be approximately one week apart
  Differences in slow oscillation-spindle coupling during non-rapid eye movement (NREM) sleep as measured by EEG between placebo and auditory stimulation naps

SECONDARY OUTCOMES:
Differences in sleep-dependent consolidation of motor procedural memory | Placebo and auditory stimulation naps will be approximately one week apart
  Differences in sleep-dependent improvement of motor procedural memory performance on the finger tapping motor sequence task (MST) between placebo and auditory stimulation naps. The MST involves pressing four numerically labeled keys on a standard keypad, repeating a 5 digit sequence as quickly and accurately as possible for 12 trials at 30 seconds each separated by 30 sec rest periods. Different sequences are employed for the placebo and stimulation visits in a counter-balanced order.
Differences in slow oscillations | Placebo and auditory stimulation naps will be approximately one week apart
  Differences in slow oscillations during non-rapid eye movement (NREM) sleep as measured by EEG between placebo and auditory stimulation naps
Differences in sleep spindles | Placebo and auditory stimulation naps will be approximately one week apart
  Differences in sleep spindles during non-rapid eye movement (NREM) sleep as measured by EEG between placebo and auditory stimulation naps

CONTACTS AND LOCATIONS:
Overall Officials: Dara Manoach, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD data.